CLINICAL TRIAL: NCT03842618
Title: The Effect of Adenotonsillectomy on Asthma Control in Preschool Children With Obstructive Sleep Apnea
Brief Title: Asthma Outcomes in Children After Adenotonsillectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Diana Shafeek Ibrahiem Ghali, the principal investigator, Assiut University
Other Study IDs: AOICAA
Record Dates: First submitted 2019-02-07; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: asthma- obstructive sleep apnea-adenotonsillectomy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to assess the effect of adenotonsillectomy on level of asthma control in preschool children with obstructive sleep apnea.

DETAILED DESCRIPTION:
Asthma is the most common chronic disease in children ,in children younger than six years it is difficult to diagnose asthma as pulmonary function tests can not be performed reliably before the age six .

Wheezing is one of the main symptoms of asthma. Young children with multiple trigger wheeze as activities ,laughing and crying are more likely to have asthma compared with episodic (viral) wheeze.

The mainstay of asthma control is daily administration of inhaled corticosteroids, long acting beta2 agonists and avoid exposure of asthma triggers as seasonal allergens and environmental pollution particularly tobacco smoke exposure.

Recent studies have found asthma to be associated with overlapping comorbidities including gastroesophageal reflux,obesity and obstructive sleep apnea.This studies have introduced therapeutic strategies aimed at improving asthma control by management of these coexisting conditions.

Pathophysiological feature of childhood obstructive sleep apnea is presence of increased airway inflammation promoting of hypertrophy of upper airway adenotonsillar tissues .

The latter promotes increased pharyngeal resistance thus predispose the upper airway to episodically collapse and cause fragmented sleep that characterize obstructive sleep apnea.

Surgically adenotonsillectomy is the first line of therapy in childhood obstructive sleep apnea and has favorable outcomes ,including improvements of respiratory sleep disturbances and in reducing markers of asthma and reduction in the use of asthma therapies.

ELIGIBILITY:
Inclusion Criteria:

* preschool children (2_5)years with criteria of bronchial asthma with obstructive sleep apnea regardless sex.

Exclusion Criteria:

* patients with other disorders that may cause obstructive sleep apnea as cranio facial syndrome , Down syndrome, cerebral palsy ,obesity,sickle cell disease, low birth weight.
* Any associated medical comorbidity that contraindicates general anesthesia.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: study will be carried out on pre school children with bronchial asthma undergoing adenoidectomy or adenotonsilectomy for obstructive sleep apnea. The study will be conducted in otolaryngology department, Assiut university hospital. The study will be carried on 60 consecutive cases.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
preschool children who suffer from bronchial asthma will be assessed by questionnaire based history to assess level of asthma control as stated in GINA 2018 before and after adenotonsillectomy. | up to 1year
  Questionnaire based history will be obtained from the parents of children before adenotonsillectomy to assess level of asthma control in preschool children as stated in Global Initiative for Asthma (GINA 2018); ask parents in the past 4 weeks, has child had A-Day time asthma symptoms for more than a few minutes, more than once a week? B-Any activity limitation due to asthma? (Runs, tires easily, playing?) C-Reliever medication needed more than once a week? D-Any night waking or night coughing due to asthma? The child will be well controlled if none of this question were answered by yes.
  The child will be partially controlled if 1-2 of this question were answered by yes.
  The child will be un controlled if 3-4 of these questions were answered by yes. Repeat this questions after adenotonsillectomy to show prognosis of asthma after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Diana shafeek Ibrahiem Ghali, Resident, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided